CLINICAL TRIAL: NCT06154928
Title: Investigation of the Effect of Drinking Warm Water on the Gastrointestinal System Functions of Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effects of Warm Water on GI System in Laparoscopic Cholecystectomy Patients
Acronym: LCSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İslam Elagöz (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Sponsor-Investigator, İslam Elagöz, Research Assıstant, Kilis 7 Aralik University
Organization: Kilis 7 Aralik University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Kilis7AralikUNİ
Record Dates: First submitted 2023-03-22; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Laparoscopic Cholecystectomy; Abdominal Distention
Keywords: Laparoscopic Cholecystectomy; Bowel Movements

STUDY DESIGN:
Intervention Model Description: This single-center randomized controlled study, conducted between January 15 and May 15, 2022, comprised 100 patients equally divided into the Water Group (WG) and Control Group (CG). Patients in the WG were allowed to take warm water orally during the 2nd postoperative hour without waiting for the onset of bowel sounds or flatus while those in the CG were not. GI functions were evaluated at 2, 4, 8, and 12 postoperative hours and the findings were recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Groups (No Intervention): Routine treatment and care of patients in the CG was continued. The onset of bowel sounds and flatus requires the initiation of oral fluid and nutrient intake. Patients in the CG were evaluated at T0, T1, T2, and T3, and data were recorded on a data collection form.
- Wather Groups (Experimental): Patients in the WG were provided warm water at the 2nd postoperative hour on the day of surgery. Patients in the WG were evaluated at T0, T1, T2, and T3 and data were recorded on a data collection form. The onset of bowel sounds and flatus requires the initiation of oral fluid and nutrient intake. No other water or food was provided to patients who had no bowel sounds or flatus other than warm water.
  Interventions: Other: Drinking Warm Water Intervention

INTERVENTIONS:
Other: Drinking Warm Water Intervention — Patients in the Warm Water Group (WG) received a warm water drinking intervention post-laparoscopic cholecystectomy. Before intake, the bed head was elevated to 45°C, and gagging and swallowing reflexes were assessed using an Abeslang to touch the oropharynx. Nausea indicated a positive reflex. Two patients with negative reflexes were excluded from WG. To maintain water temperature, individual insulated cups with thermal features were used, preventing infection transmission. Water was boiled in a clinic kettle, cooled to 37-38°C, and given to patients to drink within 15 minutes. Swallowing ability was monitored after the first sip; successful swallowing allowed the patient to continue. Patients were observed for 15 minutes with an aspirator on standby for aspiration risks. No complications occurred during the water drinking process in WG.
  Arms: Wather Groups

SUMMARY:
Objective: The study was carried out to determine the effect of drinking warm water on GIS functions in patients who underwent laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
Method: The research was completed in Kahramanmaraş Necip Fazıl City Hospital with 100 patients, 50 of whom were in the Study Group (WG) and 50 were in the Control Group (KG). The patients in CG were given warm water to drink at the 2nd hour after surgery. On the other hand, patients in KG were allowed to drink warm water after bowel sounds started and gas was produced. Patients in both groups were 2,4,8,12 after surgery. hours were evaluated in terms of GIS functions. Statistical analysis was done in SPSS 22.0 for Windows package program. A p<0.05 value was accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* having surgery

Exclusion Criteria:

* not meeting the sampling criteria
* Refused to participate Canceled surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Descriptive Information Form: | up to 18 weeks
  The descriptive information form consisted of two parts. The first part comprised seven open-ended and five multiple-choice questions to determine the patients' descriptive characteristics. This part of the form was completed by the patients 1 day before surgery. The second part comprised nine multiple-choice questions aimed at determining the patients' surgical characteristics. This diagnostic information was provided by the researcher.

SECONDARY OUTCOMES:
Postoperative Measurement and Evaluation Form: | up to 18 weeks
  The postoperative measurement and evaluation form included nine open-ended and seven multiple-choice questions designed to determine the vital signs and GI functions of the patients. Patients were evaluated during the postoperative period and the findings are presented in the relevant sections.

CONTACTS AND LOCATIONS:
Locations (1):
- Necip Fazıl Kısakürek Şehir Hastanesi, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No